CLINICAL TRIAL: NCT04231188
Title: Evaluating the User Experience of a Mobile Application in Recording Primary Caregiver Reported Outcomes of Infants
Brief Title: User Experience of a Mobile Application
Acronym: SMart
Status: Terminated | Type: Observational
Why Stopped: Delay in recruitment due to covid and a newer version of mobile app is available for testing.
Sponsor: Danone Asia Pacific Holdings Pte, Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: EBB19GC27359
Record Dates: First submitted 2019-12-06; First posted 2020-01-18 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: User Experience of Mobile Application

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Primary Caregiver and infant pair: Primary Caregiver and infant who is less than or equal to 12 months old

SUMMARY:
To evaluate the user experience of the use of the different modules / trackers in the mobile application in recording primary caregiver reported outcomes of infants

DETAILED DESCRIPTION:
Using a questionnaire to collect overall user experience, frequency of usage, feedback of each module in the mobile application

ELIGIBILITY:
Inclusion Criteria:

1. Infants from birth to ≤ 12 months of age.
2. Primary caregiver should have access to the internet and a smartphone or tablet to access the mobile application.
3. Primary caregiver should be able to comprehend the content in the mobile application and complete the questionnaires in English.
4. Primary caregiver takes care of the infant more than 50% of the time

Exclusion Criteria:

* Incapability of the primary caregiver to access the mobile application using a smartphone or tablet with internet

Max Age: 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants from birth to ≤ 12 months of age and their primary caregiver
Sampling Method: Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2019-12-26 (Actual); Primary Completion 2020-06-26 (Actual); Study Completion 2020-06-26 (Actual)

PRIMARY OUTCOMES:
Overall User experience | Day 14
  Using a questionnaire to assess primary caregiver reported overall experience on a 5-point scale (Very Poor to Very Good) of the mobile application

SECONDARY OUTCOMES:
User experience (ease of use) - Primary Caregiver | Day 14
  Using a questionnaire to assess primary caregiver ease of use (Very Poor to Very Good or Did Not Use) of use of different modules/trackers in the mobile application
User experience (frequency of use) - Primary Caregiver | Day 14
  Using a questionnaire to assess primary caregiver frequency (Rarely to Always) of use of different modules/trackers in the mobile application
User experience (usefulness) - Healthcare Professionals (HCP) | Day 14
  Using a questionnaire to assess HCP reported usefulness (not useful at all to very useful) of the data generation by the mobile application
User experience (relevance) - Healthcare Professionals (HCP) | Day 14
  Using a questionnaire to assess HCP reported relevance (not relevant at all to very relevant) of the data generation by the mobile application

OTHER OUTCOMES:
User experience (ease of use) - Primary Caregiver from Day 0 to Day 45 | Day 0 to Day 45
  Using a questionnaire to assess primary caregiver reported user experience of different modules/trackers in the mobile application on a 5-point scale (Very Poor to Very Good) of the mobile application
User experience (frequency of use) - Primary Caregiver from Day 0 to Day 45 | Day 0 to Day 45
  Using a questionnaire to assess primary caregiver reported user frequency of use of different modules/trackers in the mobile application on a 5-point scale (Rarely to Always) of the mobile application
User experience (quality of insights) - Primary Caregiver from Day 0 to Day 45 | Day 0 to Day 45
  Using a questionnaire to collect quality of insights on a 5-point scale (Very Poor to Very Good) to describe primary caregiver reported events in the modules/trackers in the mobile application
User experience (weighing scale) - Primary Caregiver from Day 0 to Day 45 | Day 0 to Day 45
  Using a questionnaire to assess primary caregiver user experience on a 5-point scale (Very Poor to Very Good) for the use of the weighing scale in measuring weight of their infants
User feedback (weighing scale) - Primary Caregiver from Day 0 to Day 45 | Day 0 to Day 45
  Using an open-ended question to collect primary caregiver feedback for the use of the weighing scale in measuring weight of their infants

CONTACTS AND LOCATIONS:
Overall Officials: Poh Choo Khoo, MBBS, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore